CLINICAL TRIAL: NCT02309606
Title: Investigation of Serotonin Receptor Binding in the Migraine Brain Using Positron Emission Tomography
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Marie Deen Christensen, Medical Doctor, Danish Headache Center
Other Study IDs: H-6-2014-057
Record Dates: First submitted 2014-12-02; First posted 2014-12-05 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Migraine without aura: Migraine patients suffering from migraine 0-4 days per month.
  Interventions: Other: PET scan with 5-HT receptor ligands
- Healthy controls: Healthy controls with no history of migraine or other primary headaches.
  Interventions: Other: PET scan with 5-HT receptor ligands
- Chronic migraine: Migraine patients with chronic migraine
  Interventions: Other: PET scan with 5-HT receptor ligands

INTERVENTIONS:
Other: PET scan with 5-HT receptor ligands — Interictal episodic migraine patients and healthy controls will be scanned with a 5-HT1B and a 5-HT4 receptor radioligand. Episodic migraine patients will further be scanned during a cilostazol induced migraine attack and after treatment with sumatriptan. Chronic migraine patients will be scanned with only the 5-HT4 receptor radioligand.

SUMMARY:
Migraine affects 16% of the world population and is one of the most disabling of all disorders. It is a complex brain disorder characterized primarily by recurrent headache attacks. The signaling molecule serotonin (5-hydroxytryptamine, 5-HT) has for decades been thought to play a central role in migraine pathophysiology. The most effective class of abortive migraine drugs, the triptans, act on 5-HT receptors. However, the migraine-specific actions of serotonin and the mechanisms of triptans are still unknown. In this project the investigators will use high-resolution positron emission tomography and specific radioligands to investigate the significance of serotonin in migraine. Two newly developed radioligands that are specific for the 5-HT1B and 5-HT4 receptor, respectively, will be applied. To investigate the level and distribution of serotonin in the migraine brain the investigators will compare the binding of these ligands in episodic migraine patients with healthy controls. In addition, the investigators will include chronic migraine patients to evaluate the relation between the level of serotonin in the brain and the frequency of migraine attacks. To investigate the changes in the serotonin level during a migraine attack and the effects of triptans on the central nervous system the investigators will repeat the scans using the 5-HT1B specific ligand during induced migraine attacks and following treatment with sumatriptan. The results from this study will shed light on the role of serotonin in the migraine brain and elucidate the migraine-specific action of triptans. This will improve our understanding of the migraine pathophysiology and, potentially, facilitate the development of more efficient treatment of migraine.

ELIGIBILITY:
Inclusion Criteria, both groups:

• Written informed consent

Inclusion Criteria, episodic migraine patients:

* Migraine without aura according to the International Headache Society (IHS) 0-4 days per month
* The migraine is treatable with sumatriptan

Inclusion Criteria, chronic migraine patients: Fulfill IHS criteria for chronic migraine

Inclusion Criteria, healthy controls:

* Do not suffer from migraine according to IHS
* Do not have any first degree relatives with migraine

Exclusion Criteria:

* Tension type headache more than 5 days per month during the last year.
* Tension type headache on the experimental day.
* Any other primary headache disorder
* Migraine 48 hour before and after the experimental day (only episodic migraine patients)
* Use of antimigraine medication or pain-killer on the experimental day before PET
* Pregnant or breastfeeding women.
* Contraindications against MRI.
* History or clinical sign of cardio- or cerebrovascular disease.
* Untreated severe mental disorder or drug abuse.
* Other diseases or disorders interpreted, by the examining doctor, to interfere with participation in the study.
* Not accepting information about potential accidental findings during the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migraine patients and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Differences in binding of the 5-HT1B radioligand | Up to 1 year
  Differences in bindingpotentials for the 5-HT1B ligand between migraine patients and healthy controls will be assessed using the Simplified Reference Tissue Model.
Differences in binding of the 5-HT4 radioligand | Up to 1 year
  Differences in bindingpotentials for the 5-HT4 ligand between migraine patients and healthy controls will be assessed using the Simplified Reference Tissue Model.
Differences in binding of the 5-HT4 radioligand | Up to 1 year
  Differences in bindingpotentials for the 5-HT4 ligand between chronic migraine patients and healthy controls and between chronic and episodic migraine patients will be assessed using the Simplified Reference Tissue Model.
Correlation with migraine frequency and 5-HT4 receptor binding | Up to 1 year
  Correlations between migraine days and 5-HT4 receptor binding will be investigated using pooled data from episodic and chronic migraine patients on migraine frequency and their 5-HT4 receptor binding potentials assessed using the simplified reference tissue model
Differences in binding of the 5-HT1B radioligand | Up to 1 year
  Differences in binding between ictal and interictal binding and between ictal and post-treatment binding in episodic migraine patients will be assessed using the simplified reference tissue model

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Hospital, Glostrup, Copenhagen, Denmark